CLINICAL TRIAL: NCT00546923
Title: A Randomized, Double-Blind, Placebo-Controlled, Pilot Study To Evaluate The Efficacy And Safety Of Venlafaxine Extended-Release In Depressed And Anxious Patients With Multiple, Unexplained Somatic Symptoms
Brief Title: Study Evaluating Venlafaxine Extended-Release in Depressed and Anxious Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0600B-101568
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2007-10

CONDITIONS: Anxiety Disorders; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

INTERVENTIONS:
Drug: Venlafaxine XR

SUMMARY:
To examine the efficacy and safety of venlafaxine XR in the treatment of physical and emotional symptoms in patients with an operationally-defined diagnosis of multisomatoform disorder (MSD).

DETAILED DESCRIPTION:
The purpose of this study is to examine the efficacy and safety of venlafaxine XR in the treatment of physical and emotional symptoms in patients with an operationally-defined diagnosis of MSD. Primary efficacy will be evaluated using the PHQ-15 scale, and secondary efficacy will be evaluated using the HAM-D17, HAM-A, CGI, MQOL-PS, VAS and SF-36 evaluation scales. Assessment scales and questionnaires will be administered at specified clinical visits between screening and Week 12 (or discontinuation).

ELIGIBILITY:
Inclusion Criteria:

· Subjects must be at least 18 years of age and meet DSM-IV diagnostic criteria for major depressive disorder, generalized anxiety disorder, and/ or social anxiety disorder, meet clinical criteria for MSD, have a total score of greater than or equal to 14 on the HAM-D17 or a total score of greater than or equal to 12 on the HAM-A at screening and no more than a 25% decrease in total HAM-D17 score or total HAM-A score from screening to randomization.

Exclusion Criteria:

* a history of an inability to tolerate or failure to respond to greater than or equal to 2 antidepressants of sufficient dose and duration of administration for the treatment of symptoms present in the current illness;
* a current or past history of mania, bipolar disorder, schizophrenia, or other psychotic disorder;
* history of seizure disorder other than childhood febrile seizure;
* presence of a serious or clinically unstable medical illness or psychiatric condition that would compromise the participation in the study;
* previous intolerance or hypersensitivity to venlafaxine or venlafaxine XR or nonresponse to a previous adequate trial of any of these drugs, or use of any nonpsychopharmacologic drug with psychotropic effects within 7 days of study randomization;
* Use of MAOI or fluoxetine within 30 days of screening; or
* Use of ECT within 3 months of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210
Dates: Start 2004-08; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change from baseline to Week 12 in the PHQ-15 total score.

SECONDARY OUTCOMES:
Efficacy will be evaluated by changes in the total scores of the HAM-D17, HAM-A, CGI, MQOL-PS, VAS and SF-36. Safety will be monitored by collecting spontaneously reported adverse events; vital signs and laboratory measures according to the Schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer